CLINICAL TRIAL: NCT05904561
Title: Effect of Low Level Laser Therapy Versus Pulsed Ultrasound on Postpartum Carpal Tunnel Syndrome
Brief Title: Effect of Low Level Laser Therapy Versus Pulsed Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mai Mahmoud Abdelmonem
Record Dates: First submitted 2023-06-01; First posted 2023-06-15 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Carpal Tunnel Syndrome; POSTPARTUM CARPAL TUNNEL SYNDROME
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (A) (Study group A) (Active Comparator): It will be consisted of 16 women complaining from mild to moderate Carpel Tunnel Syndrome after 6 weeks from delivery diagnosed by electrophysiological study. They will receive low level laser therapy, for 10 minutes, three times per week for 4 weeks (total of 12 sessions), in addition to wrist exercises and home advices.
  Interventions: Radiation: low level laser therapy
- Group (B) (study group B) (Experimental): It will be consisted of 16 women complaining from mild to moderate Carpel Tunnel Syndrome after 6 weeks from delivery diagnosed by electrophysiological study. They will receive pulsed ultrasound therapy, for 10 minutes, three times per week for 4 weeks (total of 12 sessions), in addition to wrist exercises and home advices
  Interventions: Radiation: low level laser therapy
- Group (C) (control): (Active Comparator): It will be consisted of 16 women complaining from mild to moderate Carpel Tunnel Syndrome after 6 weeks from delivery diagnosed by electrophysiological study. They will receive wrist exercises (strengthening exercises for thenar muscles, wrist flexors. Extensors, grip strengthening, stretching, nerve glide, neurodynamic technique and tendon glide) for 15 minutes, three times per week for 4 weeks (total of 12 sessions) and home advices only.
  Interventions: Radiation: low level laser therapy

INTERVENTIONS:
Radiation: low level laser therapy — comparing between the effect of low level laser therapy (LLLT) and pulsed ultrasound on post-partum carpal tunnel syndrome. All interventions that were pre-specified to be administered as part of the protocol, even if a particular intervention is not "of interest
  Other Names: pulsed ultrasound waves

SUMMARY:
Carpal tunnel syndrome (CTs), the most common entrapment neuropathy of the upper extremity, is caused by compression of the median nerve as it travels through the carpal tunnel.

CTs was clinically diagnosed in more than half of women (62%). Neurophysiological evaluation diagnosed that CTs in around half of women (43%) was positive in one hand at least, also, it was reported that about half of women with CTs during pregnancy still complained of CTs symptoms one year after delivery.

DETAILED DESCRIPTION:
Carpal tunnel syndrome pain and discomfort during postpartum period may interfere with the mother ability to successfully breastfeed due to increased physical load on the mother's hands and repetitive need for flexion during breastfeeding and carrying of the baby.

Observation of peripheral oedema in about 80% of pregnant women, especially in the period of third trimester is common, it is due to hormonal changes that cause reduction of venous return, fluid retention which decrease the carpal tunnel diameter and increase compression of the median nerve. Also, increase production of relaxin hormone leads to relaxation of the transverse carpal ligament and flattening of it that increase compression of the median nerve.

Symptoms of CTs differ from tingling, numbness and palmar side pain in radial 3.5 fingers. Typically, at night, patients are awakened by a numb hand. Complaints like decrease in hand strength, difficulty of holding things and dropping are common. Sensory distribution, median nerve hypoesthesia, positive provocative tests and atrophy or weakness of the thenar muscles may be shown in physical examination.

Nerve conduction study (NCS) has been showed as the gold standard in the diagnosis of CTs since it provides information about the physiological health of median nerve over the carpal tunnel. NCS measures sensory and motor nerve action potential which determines the severity of nerve entrapment.

Conservative treatment of CTs includes; local steroid injection, non-steroidal anti-inflammatory drugs, splinting, modification of activity, physical therapy modalities like ultrasound, low level laser therapy and stretching exercises.

Low level Laser therapy (LLLT) has analgesic and anti- inflammatory effect. Also, LLL improves the metabolic processes and increases protein synthesis that improves blood flow, blood vessel health and cell regeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Postpartum women with mild to moderate carpal tunnel syndrome will participate in this study.
2. Their ages will range from 25 to 35 years old.
3. Their BMI will be ranged from 25 to 30 Kg/m2.
4. The electrophysiological evidence of mild or moderate median nerve lesion at wrist (mild: sensory nerve conduction velocity slow on finger/wrist measurement, sensory nerve latency >3.5 ms, normal terminal motor latency; moderate: sensory potential preserved with motor slowing, distal motor latency to abductor pollicis brevis (APB) < 6.5 ms) (Bland, 2000 and Dumitru and Zwarts, 2002).
5. Positive phalen's test.
6. Positive tinel's test.
7. Unilateral or bilateral carpal tunnel affection will be included.

Exclusion Criteria:

1. History of brachial plexopathy or malignancy.
2. Radial, ulnar neuropathy, proximal median neuropathy or polyneuropathy.
3. Previous wrist surgery or steroid injection for carpal tunnel syndrome.
4. History of trauma, fracture, deformity or inflammation in the wrist, such as rheumatoid arthritis.
5. Coagulation abnormalities, pregnancy, fever and infections.
6. Skin disease and skin cancer.
7. Spots, birthmarks or tattoos over the work points.
8. Pacemaker and implementable medical devices.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | From base line to 4 weeks from starting the treatment
  measure pain intensity for each woman in all groups (A, B and C). The VAS is usually presented as a 10-cm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable." Its simplicity, reliability and validity, as well as its ratio scale properties make the VAS the optimal tool for describing pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Afaf Mohammed, Assist.Prof., Study Chair — Department of physical Therapy for Women's Health, Faculty of Physical Therapy Cairo University
Locations (1):
- Faculty of Physical Therapy - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided